CLINICAL TRIAL: NCT02096510
Title: Ultradian Subcutaneous Hydrocortisone Infusion in Addison Disease and Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013/1738
Record Dates: First submitted 2013-11-28; First posted 2014-03-26 (Estimated); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Addison Disease; Adrenal Hyperplasia Congenital
Keywords: Addison Disease; Adrenal Hyperplasia Congenital
MeSH Terms: conditions — Addison Disease; Adrenal Hyperplasia, Congenital | interventions — hydrocortisone hemisuccinate; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- continuous subcutaneous hydrocortisone (Experimental): continuous subcutaneous hydrocortisone infusion (CSHI), Solu-Cortef ® 50mg/ml infusate
  Interventions: Drug: Solu-Cortef; Drug: Cortef
- cortef tablets (Active Comparator): the patient regular treatment by Cortef 5 mg, produced by Nycomed Pharma two times or three times a day.
  Interventions: Drug: Solu-Cortef; Drug: Cortef
- ultradian subcutaneous hydrocortisone (Experimental): ultradian subcutaneous hydrocortisone infusion, Solu-Cortef ® 50mg/ml infusate
  Interventions: Drug: Solu-Cortef; Drug: Cortef

INTERVENTIONS:
Drug: Solu-Cortef — administration by pump for minimum 2 weeks
  Other Names: hydrocortisone
Drug: Cortef — tablet treatment 2 ro 3 times per day for 14 days
  Other Names: hydrocortisone tablets

SUMMARY:
The aim of this study is to compare the effects of tablet treatment, circadian and combined circadian and ultradian subcutaneous hydrocortisone infusion on steroid metabolism and tissue responses to therapy.

DETAILED DESCRIPTION:
The conventional glucocorticoid replacement therapy in primary adrenal insufficiency (Addison's disease) and congenital adrenal hyperplasia renders the cortisol levels unphysiological, which may cause symptoms and long-term complications. This therapeutical approach does not enable to restore physiological circadian and ultradian rhythm of glucocorticoids. Current studies conclude that constant or unphysiological administration of glucocorticoids leads to abnormal gene transcription and causes sides effect of glucocorticoids treatment and long standing complications Glucocorticoid replacement is technically feasible by continuous subcutaneous hydrocortisone infusion, which can mimic not only the normal diurnal cortisol rhythm, but potentially also the ultradian cadence.

This is a pilot trial with an open cross-over design of 3 x minimum 2 weeks in 10 patients comparing the effects of tablet treatment versus continuous subcutaneous hydrocortisone infusion versus ultradian subcutaneous hydrocortisone infusion on serum, salivary, tissue hormonal response and glucocorticoid related gene expression.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of primary adrenal insufficiency
2. Written informed consent

Exclusion Criteria:.

1. Diabetes mellitus
2. Severe cardiovascular disease
3. Active malignant disease
4. Pregnancy or breast feeding
5. treatment with interfering drugs
6. Intake of grapefruit juice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Serum cortisol -24 hours curve | 24 hours
  admission to hospital for 24 hours

SECONDARY OUTCOMES:
Salivary cortisol - 24 hours curve | 24 hours
  admission to the hospital for 25 hours
24 h urine cortisol and metabolites | 24 hours
  urine samples for 24 hours
levels of corticotropic hormone | 24 hours
  blood samples
24 hours curve of tissue cortisol | 24 hours
  The tissue effect of glucocorticoid replacement - 24 hours curve of tissue cortisol (microdialysis)
gene expression | 24 hours
  m RNA expression of genes

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Simunkova, MD, PhD, Principal Investigator — Universtity of Bergen; Kristian Løvås, MD, PhD, Study Director — Helse Bergen
Locations (1):
- University Hospital Helse Bergen, Bergen, Norway

REFERENCES:
- [Background] Lightman SL, Conway-Campbell BL. The crucial role of pulsatile activity of the HPA axis for continuous dynamic equilibration. Nat Rev Neurosci. 2010 Oct;11(10):710-8. doi: 10.1038/nrn2914. Epub 2010 Sep 15. PMID 20842176
- [Background] Lovas K, Husebye ES. Continuous subcutaneous hydrocortisone infusion in Addison's disease. Eur J Endocrinol. 2007 Jul;157(1):109-12. doi: 10.1530/EJE-07-0052. PMID 17609409
- [Background] Lightman SL, Windle RJ, Julian MD, Harbuz MS, Shanks N, Wood SA, Kershaw YM, Ingram CD. Significance of pulsatility in the HPA axis. Novartis Found Symp. 2000;227:244-57; discussion 257-60. doi: 10.1002/0470870796.ch14. PMID 10752074
- [Result] Simunkova K, Lovas K, Methlie P, Jovanovic N, Bifulco E, Bronstad I, Lightman SL, Husebye ES, Oksnes M. Pulsatile Subcutaneous Hydrocortisone Replacement in Primary Adrenal Insufficiency. Horm Metab Res. 2023 Jul;55(7):471-478. doi: 10.1055/a-2092-5228. Epub 2023 May 12. PMID 37172949